CLINICAL TRIAL: NCT02386046
Title: Does the Use of Caffeine Post Discharge Normalize the Respiratory Patterns in Infants Born Earlier Than 35 Weeks? A Cohort Study
Brief Title: Oxygen Saturation and Caffeine Post-Discharge
Acronym: OCPDPS
Status: Terminated | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Carlos Fajardo, Clinical Associate Professor, University of Calgary
Other Study IDs: REB14-0175
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2017-05

CONDITIONS: Prematurity
Keywords: Caffeine use; Normative data
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reference Group: Late preterm infants without any pathology. Intervention: Pulse oxymeter measurements at the hospital and weekly thereafter until 46 weeks postconceptional age.
  Interventions: Other: Pulse oxymeter measurements
- Study Group: Infants born 26-35 weeks requiring caffeine. Intervention: Pulse oxymeter measurements at the hospital before and after caffeine instituted, and weekly thereafter until 46 weeks postconceptional age.
  Interventions: Other: Pulse oxymeter measurements
- Control Group: Infants born 26-35 weeks not requiring caffeine. Intervention: Pulse oxymeter measurements at the hospital and weekly thereafter until 46 weeks postconceptional age.
  Interventions: Other: Pulse oxymeter measurements

INTERVENTIONS:
Other: Pulse oxymeter measurements — Pulse oxymeter measurements done at the hospital and upon discharge, weekly until 46 weeks postconceptional age

SUMMARY:
This study aims to determine normative values of oxygen saturation in late preterm infants, and evaluate the frequency of hypoxic events in infants requiring caffeine at discharge and those not requiring it.

DETAILED DESCRIPTION:
Apnea of prematurity is a common morbidity among premature infants. Recent studies suggest an association between apnea and neurodevelopmental impairment. Our objectives are to determine normative values of oxygen saturation in late preterm infants -reference group. In infants born 28-35 weeks requiring caffeine- study group and infants born 28-35 weeks not requiring caffeine-control group we will be evaluating the frequency of hypoxic events. Recruitment time: February 2015 until December 2016.

After consent a pulse oxymeter will be placed on the infant's right wrist. For those infants that will receive caffeine prior to discharge, this medication will be instituted after 12 hours of the initiation of the study and continue for the remaining of the hospitalization. For all other infants, the pulse oxymeter will be done continuously until discharge. After discharge, the recording will be done at home once a week until 46 weeks corrected age in the three groups.

All the data will be reviewed by a blind observer to the groups from which that data comes. The data will be analyzed by a statistician.

Normative values will be developed on the reference group until 46 weeks post conceptional age.

Any medical problems encounter by the patients while on the study or in the following 6 months will be recorded to establish the safety of caffeine use at home and its discontinuation at 44 weeks post conceptional age.

ELIGIBILITY:
Inclusion Criteria of infants admitted to NICU:

1. Gestational age at birth of < or = 35 weeks
2. Families of infants that live in Calgary
3. Infants discharged home from PLC or South Health Campus (SHC)
4. Decision of treating team to start caffeine
5. No episodes of clinically significant apnea for a period of 3 to 5 days prior to discharge
6. Infant has access to reliable post-discharge follow up

Exclusion Criteria of all infants:

1. Active serious medical conditions other than apnea (Congenital Heart Disease (CHD), Chronic Lung Disease (CLD), symptomatic anemia).
2. Congenital disorders like Trisomies, genetic syndromes, midline defects, metabolic disorders.

Ages: 26 Weeks to 46 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants admitted at two NICU centers in Calgary born prematurely between 26 weeks and 34 weeks of gestational age.
  Newborn infants admitted directly to the normal nursery in those two centers born less than 38 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Pattern of Oxygen saturation | Up to 46 weeks postconceptional age
  Measurements at hospital and weekly after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Fajardo, Md, Principal Investigator — University of Calgary; Veronica Samedi, Md, Study Director — Alberta Health services
Locations (1):
- Peter Logheed Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided